CLINICAL TRIAL: NCT04614792
Title: Excitatory Prefrontal Weak Current Stimulation in Vegetative Patients:Potential to Induce Modulation in Neurocognitive Features of Awareness
Brief Title: Excitatory Prefrontal Weak Current Stimulation in Vegetative Patients
Acronym: VEG-TDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oded Meiron (Other)
Collaborators: Neurosteer Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Oded Meiron, Director of Non-invasive Brain Stimulation Center, Herzog Hospital
Organization: Herzog Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 335-19
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Disorder of Consciousness; MMN; Modification of Cognitive Status Indication; Anoxic Brain Damage; Trauma, Brain; Vegetative State; EEG; Paroxysms, Occipital, Epilepsy of Childhood; Cortical Atrophy
MeSH Terms: conditions — Consciousness Disorders; Hypoxia, Brain; Brain Injuries, Traumatic; Persistent Vegetative State | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: open lable treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active treatment (Experimental): open label experimental treatment
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Non-invasive brain stimulation or neuromodulation.

SUMMARY:
In response to "conscious" EEG findings related to detectable cognitive function that reliably denote awareness in vegetative state patients, in the current study, we will assess the covert conscious EEG activity (as well as standard clinical overt measures) and neuroplasctic propensity (i.e., changes in EEG spectral power synchronization values following tDCS intervention) in vegetative-state patients receiving repetitive transcranial direct current stimulation (tDCS) treatment over frontal motor areas for a period of two weeks. In support of this approach, a recent tDCS study with vegetative and minimally conscious patients implied that a twenty minutes anodal stimulation (i.e., excitatory stimulation) to the left dorsolateral prefrontal cortex (DLPFC) significantly increased CRS-R scores versus sham (placebo: non-active stimulation) stimulation condition. It was noted that this tDCS effect was more pronounced in minimally conscious state patients versus vegetative state patients excluding effects of chronicity or etiology. Thus, the investigators in this study suggested that tDCS could be effective in improving cognitive recovery in severely brain-injured patients. However, their findings would benefit neural activation correlates that could support their conclusion regarding the effectiveness of this type of non-invasive intervention in promoting neurocognitive recovery. Most importantly, tDCS is safe for use in humans, has no adverse effects, is considered the most non-invasive transcranial stimulation method because it uses extremely weak currents (0.5 to 2 mA), and, is known to only temporarily shift the neuron's membrane potential towards excitation/inhibition. In regard to the method's potential to induce functional recovery in vegetative state patients, recent clinical studies indicate that tDCS could counteract the negative effects of brain damage by influencing neurophysiological mechanisms, and is likely to contribute to the "formation of functionally meaningful connections and the maintenance of existing pathways" .

ELIGIBILITY:
Inclusion Criteria:

* Anoxic brain damage/TBI/CVA/progressive dementia/encephalopathy
* Vegetative state patients or minimally conscious state according to CRS-R criteria
* Ages 18 to 90
* Consent for participation in clinical study (e.g., informed consent) by legal guardian of patients.

Exclusion Criteria:

* Intracranial metal implants
* Implanted devices that may be affected by tDCS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Active medical condition that would preclude medical stability for the study, including significant ECG abnormalities, cardiac arrhythmia, uncontrolled high blood pressure
* Participation in other research studies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
JFK COMA RECOVERY SCALE - REVISED | 24 months
  JFK Coma recovery Scale - Revised scores for diagnosing disorders of consciousness. This cynical assessment scale examines reflexive behaviors such as response to pain and startle, and touch. The CRS consists of 25 hierarchically arranged items that comprise 6 subscales addressing auditory, visual, motor, oro- motor, communication, and arousal processes. Scoring is based on the presence or absence of specific behavioral responses to sensory stimuli administered in a standardized manner. The lowest item on each subscale represents reflexive activity, whereas the highest items represent cognitively mediated behaviors. sub scales represent motor function, auditory function, visual function sub scales and arousal sub scales. The low scores indicate low levels of functioning and the higher score indicate high levels of function an awareness. Maximum score is 23 and a minimal score is 0.

SECONDARY OUTCOMES:
MMN ERP amplitudes | 2 weeks
  Prefronal-Temopral cortex neuroplasticity and reactivity to sound : size of early auditory processing ERP amplitudes. If the negative change in ERP amplitudes is larger than in indicates better change-detection and neurplasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Efraim Jaul, MD, Principal Investigator — Herzog Medical Center
Locations (1):
- Herzog Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
Treatment methods and diagnostic methods will be shared as well as change in clinical and neurological status via research publication.

REFERENCES:
- [Background] Angelakis E, Liouta E, Andreadis N, Korfias S, Ktonas P, Stranjalis G, Sakas DE. Transcranial direct current stimulation effects in disorders of consciousness. Arch Phys Med Rehabil. 2014 Feb;95(2):283-9. doi: 10.1016/j.apmr.2013.09.002. Epub 2013 Sep 11. PMID 24035769